CLINICAL TRIAL: NCT01970462
Title: Use of Sitagliptin for Stress Hyperglycemia or Mild Diabetes Following Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment
Sponsor: Kathleen Dungan (Other)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013H0328
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Patients will receive Sitagliptin (renally dosed) prior to hospital discharge and 6 weeks following discharge
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Patients will receive placebo prior to discharge and 6 weeks after discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin prior to hospital discharge and 6 weeks following discharge.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Patients are reandomized to Sitagliptin or placebo for 6 weeks post-operatively
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial to determine the safety and efficacy of Sitagliptin in patients with stress hyperglycemia or mild diabetes following cardiac surgery. Patients will receive Sitagliptin or placebo. Sitagliptin may be of particular use in this patient population due to the effects on hepatic glucose production (a major feature of SH), safety (lack of contra-indications for heart failure or renal failure and no hypoglycemia), and tolerability. The secondary objective of this study is to determine whether the management of patients with persistent insulin requirements following cardiac surgery differs among patients with stress hyperglycemia or mild diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Either of the following: Mild Diabetes Mellitus or Stress Hyperglycemia
* AND:
* Cardiac Surgery
* Insulin Requirement between 8-30 units subcutaneous on post-op day 3 or later off pressors, off enteral feeding, extubated OR glucose >150 mg/dL at least twice in a 24 hour period (>4 hours apart) and otherwise not requiring basal insulin

Exclusion Criteria:

* use of pressors, mechanical ventilation, or enteral or parenteral feeding within previous 12 hours
* glucocorticoids in doses exceeding the equivalent of Prednisone 10 mg/day within the previous 48 hours
* left ventricular assist device
* percutaneous or laparoscopic surgery
* end stage renal disease
* end stage liver disease
* history of pancreatitis
* type 1 diabetes
* pregnancy
* unable to give consent in english
* no phone
* prisoners
* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, MPH, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled differs from reported because the study was discontinued early and the group number was not available from the pharmacy for 3 subjects. We provided the participant flow for the 5 individuals for whom the group assignment was available. Of 8 total patients enrolled, 4 completed the study, 3 of whom had group assignments available
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 1 | 4
Completed | 1 | 2
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Number of patients with at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Fasting Glucose
Description: Difference in mean fasting glucose at 6 weeks post-discharge.
Time Frame: 6 weeks
Population: The study was discontinued early and the group assignment was not available from the pharmacy for 3 subjects. Therefore we are unable to provide group level data for the outcomes. Among the 4 subjects for whom data was available, the fasting 6 week glucose value was 158, 114, 83, 237 mg/dl.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Self Monitored Blood Glucose
Description: Mean blood glucose at week 2
Time Frame: 2 weeks
Population: The study was discontinued early and the group assignment was not available from the pharmacy for 3 subjects. therefore we are unable to provide group level data for the outcomes. Among the 5 subjects for whom data were available the value was 130, 134.6, 96.5, 132, 98 mg/dl
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Adherence
Description: adherence defined as 80% of all Sitagliptin doses respectively taken in previous week
Time Frame: 6 weeks
Population: The study was discontinued early and the group assignment was not available from the pharmacy for 3 subjects. therefore we are unable to provide group level data for the outcomes. Among the 5 subjects for whom data were available, 100% were adherent.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Hypoglycemia
Description: Number of subjects with glucose <70 mg/dl following time of discharge to 6 weeks.
Time Frame: 6 weeks
Population: The study was discontinued early and the group assignment was not available from the pharmacy for 3 subjects. therefore we are unable to provide group level data for the outcomes. There was no hypoglycemia reported in any of the 5 subjects for whom data were available at the 6 week timepoint.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes